CLINICAL TRIAL: NCT05732766
Title: A Phase III Randomized, Modified Double-blind, Multi-centric, Comparative Study, to Evaluate Non-inferiority, Immunogenicity and Safety Cholera Vaccine Hillchol® (BBV131) to the Comparator Vaccine Shanchol™ and Hillchol® Lot Consistency
Brief Title: To Evaluate Safety of Oral Cholera Vaccine Hillchol® (BBV131)
Acronym: Hillchol131
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Hillchol®(BBV131) Safety
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-I (Age: ≥18) (Experimental): Group-I (Age: ≥18) In this group, a total of 600 participants aged ≥18 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14.
  Interventions: Biological: Hillchol vaccine
- Group-II (Age: ≥5 to <18) (Experimental): Group-II (Age: ≥5 to <18): In this group, a total of 600 participants aged ≥5 to <18 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14.
  Interventions: Biological: Hillchol vaccine
- Group-III (Age: ≥1 to <5) (Experimental): Group-III (Age: ≥1 to <5): In this group, a total of 600 participants aged ≥1 to <5 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14
  Interventions: Biological: Hillchol vaccine

INTERVENTIONS:
Biological: Hillchol vaccine — Hillchol® (BBV131) (The whole cell inactivated Stable Hikojima expressing both Inaba and Ogawa LPS) inactivated bacteria of a stable recombinant Vibrio cholerae O1 El Tor Hikojima serotype strain expressing approximately 50% each of Ogawa and Inaba O1 LPS antigens.

SUMMARY:
A Phase III randomized, modified double-blind, multi-centric, comparative study, to evaluate the non-inferiority of immunogenicity and safety of single strain oral cholera vaccine Hillchol® (BBV131) to the comparator vaccine Shanchol™ along with lot-to-lot consistency of Hillchol®(BBV131).

Study Population: A total of 1800 participants will be enrolled in three descending age groups(Group I- ≥18, Group II: ≥5 to <18 and Group III: ≥1 to <5). In each group,600 participants will be enrolled and will receive two doses of Hillchol® (BBV131) vaccine two weeks apart.

DETAILED DESCRIPTION:
A Phase III randomized, modified double-blind, multi-centric, comparative study, to evaluate the non-inferiority of immunogenicity and safety of single strain oral cholera vaccine Hillchol® (BBV131) to the comparator vaccine Shanchol™ along with lot-to-lot consistency of Hillchol®(BBV131).

Study Population: A total of 1800 participants will be enrolled in three descending age groups(Group I- ≥18, Group II: ≥5 to <18 and Group III: ≥1 to <5). In each group,600 participants will be enrolled and will receive two doses of Hillchol® (BBV131) vaccine two weeks apart.

Study Objectives:

Primary Objectives:

1)To evaluate the frequency and severity of all solicited and unsolicited adverse events after administration of two doses of Hillchol® (BBV131) among all three age groups.

End points:

1. Immediate reaction: Within 30mins of administration of each dose.
2. Incidence, intensity, and the causality of all solicited adverse events during the 7-day follow up period after each dose.
3. Incidence, intensity, and the causality of unsolicited adverse events during the 7-day follow up period after each dose.
4. Incidence, intensity, and the causality of all adverse events and Serious Adverse Events (SAEs) during the entire study period.

Study design:

In this study, a total sample size of 1800 participants will be enrolled in three age groups and administered with Hillchol® (BBV131).

A) Group-I (Age: ≥18): In this group, a total of 600 participants aged ≥18 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14.

B) Group-II (Age: ≥5 to <18): In this group, a total of 600 participants aged ≥5 to <18 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14.

C)Group-III (Age: ≥1 to <5): In this group, a total of 600 participants aged ≥1 to <5 will be enrolled and administered two doses of Hillchol® (BBV131) on day 0 and 14.

Eligibility Criteria:

Inclusion Criteria:

1. Participants /Legally acceptable representatives who have the ability to provide written informed consent.
2. Participants of either gender of age ≥ 1 year.
3. Expressed interest and availability to fulfill the study requirements.

   1. Willing to receive two doses of the vaccine at the specific study site.
   2. Willing to be contacted on the phone to assess adverse events and for study reminders.
4. Agrees not to participate in another clinical study at any time during the study period.

Exclusion:

1. Any history of anaphylaxis in relation to vaccination.
2. Participants with Immune function disorders including immunodeficiency diseases, or taking immunosuppressive/cytotoxic agents.
3. An individual is thought to have difficulty participating in the study due to severe chronic diseases, based on the judgment of the investigator.
4. Participants with 38℃ or higher body temperature measured within 24 hours or at the time of investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours before study initiation.
6. Diarrhea or administration of anti-diarrheal drugs or antibiotics to treat diarrhea within 1 week before study initiation.
7. Other vaccination within 4 weeks before study initiation.
8. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months before study initiation.
9. Participation in another clinical trial.
10. History of cholera vaccinations or history of cholera diarrhea.
11. Pregnancy, lactation or willingness/intention to become pregnant during the study.
12. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
13. History of any psychiatric condition likely to affect participation in the study.
14. Suspected or known current alcohol abuse is defined by an alcohol intake of greater than 42 units every week.
15. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the study or would render the subject unable to comply with the protocol.

Study Procedure:

Visit 1:Baseline (Day 0):If eligible, study participants will attend the OPD for a physical and general examination. A study vaccine will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes to record any adverse events. Diary cards will be distributed to all the participants to record the adverse events after vaccination.

Day 1-7: The study participants will be telephonically followed up by the site for the first 7 days to know their current health status

. Visit 2 (Day 14+2):Study participants will return to the OPD for physical, and general examination. A study vaccine will be administered. Following vaccination, participants will remain at the study site for at least 30 minutes to record any adverse events. Diary cards will be distributed to all the participants to record the adverse events after vaccination.

Day 15-21: The study participants will be telephonically followed up by the site for the first 7 days to know their current health status.

Visit 3 (Day 28+2):Study participants will return to the OPD for physical and general examination. Diary cards will be collected from all the participants to record the adverse events after vaccination.

Visit 4: (Day 56±7):Study participants will be contacted telephonically and followed up by the site to know their current health status and all the safety-related issues will be recorded.

Visit 5 (Day 90±7):-Study participants will return to the OPD for physical and general examination. If any adverse events it will be recorded.

Visit 6 (Day 180±7):Study participants will be contacted telephonically and followed up by the site to know their current health status and all the safety-related issues will be recorded.

Unscheduled visits:

If any subject develops any adverse or serious adverse event or is concerned about his/her health, they will be advised to visit the study site during the study follow-up period. All unscheduled visits and details of adverse events will be documented in the source document. Concomitant medications, if any, will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Participants /Legally acceptable representatives who have the ability to provide written informed consent.
2. Participants of either gender of age > 1 year.
3. Expressed interest and availability to fulfill the study requirements.

   1. Willing to receive two doses of the vaccine at the specific study site.
   2. Willing to be contacted on the phone to assess adverse events and for study reminders.
4. Agrees not to participate in another clinical study at any time during the study period.

Exclusion Criteria:

1. Any history of anaphylaxis in relation to vaccination.
2. Participants with Immune function disorders including immunodeficiency diseases, or taking immunosuppressive/cytotoxic agents.
3. An individual is thought to have difficulty participating in the study due to severe chronic diseases, based on the judgment of the investigator.
4. Participants with 38℃ or higher body temperature measured within 24 hours or at the time of investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours before study initiation
6. Diarrhea or administration of anti-diarrheal drugs or antibiotics to treat diarrhea within 1 week before study initiation.
7. Other vaccination within 4 weeks before study initiation.
8. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months before study initiation.
9. Participation in another clinical trial.
10. History of cholera vaccinations or history of cholera diarrhea.
11. Pregnancy, lactation or willingness/intention to become pregnant during the study.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Immediate reaction | Within 30 mins of administration of each dose
  Adverse reactions after administration of each dose
solicited adverse events | 7-days
  Incidence, intensity, and the causality of all solicited adverse events during the 7-day follow up period after each dose.
unsolicited adverse events | 7-days
  Incidence, intensity, and the causality of unsolicited adverse events during the 7-day followup period after each dose.
Serious Adverse Events (SAEs) | V- :1Baseline (Day 0),V- 2: (Day 14+2),V-3: (Day 28+2),V- 4: (Day 56±7),V-5: (Day 90±7) and V- 6: (Day 180±7)
  Incidence, intensity, and the causality of all adverse events and Serious Adverse Events (SAEs) during the entire study period.

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - King George Hospital, Visakhapatnam, Visakhapatnam, Andhra Pradesh
  - Rajarajeswari Medical College and Hospital, Kambīpura, Bangalore
  - All India Institute of Medical Sciences, Patna, Patna, Bihar
  - Pt BD Sharma,PGIMS/UHS. Rohtak, Rohtak, Haryana
  - Jeevan Rekha Hospital, Belgaum, Belagavi, Karnataka
  - Gillurkar Multispecialty Hospital, Nagpur, Maharashtra
  - Malla Reddy Narayana Multi Speciality Hospital, Hyderabad, Telangana
  - Rana Hospital Pvt Ltd, Gorakhpur, Uttar Pradesh
  - New Leelamani Hospital Pvt Ltd, Kanpur, Uttar Pradesh